CLINICAL TRIAL: NCT06521619
Title: Analysis of Postoperative Analgesic Effect and Complications Among Different Approaches of Nerve Block for Total Knee Replacement Surgery
Brief Title: Analysis of Postoperative Analgesic of Different Nerve Blocks for Total Knee Replacement Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Principal Investigator, Sung, Chao-Hsien, Attending anesthesiologists, Fu Jen Catholic University Hospital
Other Study IDs: FJUH113365
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Pain; Total Knee Replacement; Motor Function
Keywords: Analgesia; Nerve block; Total knee replacement
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient receiving Sciatic and Femoral nerve blocks: Patient receiving Sciatic and Femoral nerve blocks
  Interventions: Procedure: Femoral and sciatic nerve blocks
- Patient receiving Adductor canal block and infiltration of posterior capsule of knee: Patient receiving Adductor canal block and infiltration of posterior capsule of knee

INTERVENTIONS:
Procedure: Femoral and sciatic nerve blocks — Patients receiving Adductor canal block and infiltration of posterior capsule of knee
  Other Names: Adductor canal block and infiltration of posterior capsule of knee
  Groups: Patient receiving Sciatic and Femoral nerve blocks

SUMMARY:
This study is a retrospective analysis using the accumulated clinical database from 2017/09-2023/11 to analyze patients who underwent total knee arthroplasty and received nerve blocks. The aim is to compare the analgesic effects, incidence of nerve injury, and rate of chronic pain under different nerve block techniques.

DETAILED DESCRIPTION:
Protocol title： Analysis of postoperative analgesic effect and complications among different approaches of nerve block for total knee replacement surgery Objectives： There is no consensus on the optimal nerve block choice for knee joint replacement. Therefore, the aim of this study is to conduct a retrospective analysis using data from patients who underwent total knee replacement (TKR) and received nerve blocks at our hospital. This study will investigate the postoperative analgesic consumption, duration of pain relief, motor function block, complications, and patient satisfaction for different nerve block techniques. The goal of this project is to identify the optimal nerve block choice to benefit future patients undergoing knee joint replacement.

Background： After undergoing total knee replacement (TKR), patients need rehabilitation to restore knee function and reduce postoperative adhesions. However, pain often prevents them from achieving this goal. Clinically, nerve block anesthesia is gradually becoming mainstream, as it achieves intraoperative anesthesia and postoperative analgesia by infiltrating local anesthetics into the nerves supplying the knee joint. According to a study by Allen et al. (1998), patients receiving nerve blocks such as femoral and sciatic nerve blocks experienced better pain relief within the first 8 hours postoperatively and had a 50% reduction in total morphine consumption on the second postoperative day compared to those who received spinal anesthesia alone. Carli et al. (2010) found that patients who received femoral nerve blocks used less postoperative patient-controlled analgesia (PCA) and had better postoperative motor function recovery compared to those who received periarticular anesthetic infiltration.

Currently, there are various types of nerve block techniques, including femoral nerve, obturator nerve, adductor canal nerve, and sciatic nerve blocks. Different nerve block techniques result in varying analgesic efficacy, duration, functional impact, motor block, and complications. Sharma et al. (2010) indicated that femoral nerve blocks might cause quadriceps muscle weakness and patient falls. Kinghorn et al. (2012) also reported that sciatic nerve blocks might result in foot drop.

Study Design： This study is a retrospective analysis using the accumulated clinical database from 2017/09-2023/11 to analyze patients who underwent total knee arthroplasty and received nerve blocks. The aim is to compare the analgesic effects, incidence of nerve injury, and rate of chronic pain under different nerve block techniques.

Methods： A. Evaluation Methods: Data is collected in a patient registry called "acute pain service" (APS), which is the medical record for documenting the dose of patient controlled analgesia and side effects of PCA or nerve blocks.

1. Duration of Pain Relief: Ask patients when they started to feel pain (duration).
2. Quantitative Assessment of Analgesic Effectiveness: Patients receiving nerve blocks will also use intra-venous patient-controlled analgesia (PCA) for 2 days postoperatively. The total amount of medication used in the PCA machine over these 2 days will reflect the patient's pain level.

i. Pain: VAS score ii. Motor Block Assessment: The motor function of patients who received nerve blocks will be evaluated for abnormalities the day after surgery. Motor block will be assessed using the Modified Bromage Motor Blockade Score. c. Complication Statistics: Defined as conditions like foot drop, quadriceps muscle weakness, or any situation requiring special medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving general anesthesia combined with nerve blocks for total knee replacement

Exclusion Criteria:

* Age less than 20 years old
* Not receiving nerve blocks
* American society of anesthesiologist physical status class greater than 4
* Contraindicated to receiving nerve blocks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Patient receiving general anesthesia combined with nerve blocks for total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain | Postoperative day 0,1,2
  Acute postoperative pain

SECONDARY OUTCOMES:
Range of motion | Postoperative day 0,1,2
  Knee passive range of motion
Analgesic consumption | Postoperative day 0,1,2
  PCA dose consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No
Patient data is protected under privacy guidelines of our institute and the need of original patient data could be obtained by written mail request to study officials and the request would be reviewed by our institute.

REFERENCES:
- [Derived] Sung CH, Liu JH, Hung CF, Fu CH. Comparative analysis of adductor canal block combined with iPACK block versus femoral combined with sciatic nerve blocks: a propensity score matched study. BMC Anesthesiol. 2025 May 16;25(1):249. doi: 10.1186/s12871-025-03112-z. PMID 40380131